CLINICAL TRIAL: NCT03197922
Title: A Multidisciplinary Approach to the Treatment of Encopresis in Children With Autism Spectrum Disorders
Brief Title: Treatment of Encopresis in Children With Autism Spectrum Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nathan A. Call, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00095849
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Encopresis; Autism Spectrum Disorder
Keywords: Constipation
MeSH Terms: conditions — Encopresis; Autism Spectrum Disorder; Constipation | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 56 participants will be assigned to 2 weeks of the Multidisciplinary Intervention for Encopresis (MIE) treatment, 56 will be assigned to treatment as usual (TAU) as a control group. Twenty-six participants were assigned to the study arm with one week of MIE, which has been discontinued.
Who Masked: Outcomes Assessor
Masking Description: Outcome measures, including the Parent-nominated Target Problem (PTP), will be conducted by separate independent evaluators (IE) each of who are blind to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MIE Treatment for Two Weeks (Experimental): Participants in this arm will receive the Multidisciplinary Intervention for Encopresis (MIE) for two weeks. MIE consists of daily clinic appointments, each of which lasts until a continent bowel movement occurs or 3 hours elapse. These participants will discontinue the use of medication previously prescribed for the treatment of constipation, other than the suppositories used in the MIE treatment. During MIE, medical professionals resolve any constipation and oversee a regimen of over the counter medications that increase the predictability of a bowel movement.
  Interventions: Behavioral: MIE Treatment; Drug: Glycerin Suppository
- Treatment as Usual (TAU) (Active Comparator): Participants randomized to the Treatment as Usual (TAU) group will continue to receive outpatient medical treatment of encopresis according to best practice guidelines by the pediatric gastroenterologist. Additionally, participants in the TAU group will receive a 2-hour long individual appointment with a doctoral level clinician with extensive experience in behavioral treatments for encopresis.
  Interventions: Combination Product: Treatment as Usual (TAU)
- MIE Treatment for One Week (Experimental): Participants in this arm will receive the Multidisciplinary Intervention for Encopresis (MIE) for one week. This study arm was discontinued in October 2019.
  Interventions: Behavioral: MIE Treatment; Drug: Glycerin Suppository

INTERVENTIONS:
Behavioral: MIE Treatment — Appointments consist of a series of sitting routines (i.e., "sits"). Each sit consists of 10 min on the toilet, followed by 1 min of standing, then repeating the 10 min on the toilet 1 min off, for up to 32 cumulative minutes of sitting. The first sit occurs prior to the administration of any medication providing an opportunity for an independent continent bowel movement.
  Other Names: Multidisciplinary Intervention for Encopresis
  Arms: MIE Treatment for One Week; MIE Treatment for Two Weeks
Drug: Glycerin Suppository — If no continent bowel movement occurs with the first sit, trained staff administer a dose of a liquid glycerin suppository, immediately followed by another sit to ensure any resulting bowel movement is continent. Glycerin suppositories are replaced by bisacodyl if 2 days pass without a continent bowel movement using the liquid glycerin suppository. Behavioral intervention consists of potent positive reinforcers when a continent bowel movement occurs. As independent continent bowel movements begin to occur, the need for the medical regimen diminishes, and is gradually faded out entirely.
  Arms: MIE Treatment for One Week; MIE Treatment for Two Weeks
Combination Product: Treatment as Usual (TAU) — Participants randomized to the Treatment as Usual (TAU) group will continue to receive outpatient medical treatment of encopresis according to best practice guidelines by the pediatric gastroenterologist. In addition, participants in the TAU group will receive a 2-hour individual appointment in clinic with a doctoral level clinician with extensive experience in behavioral treatments for encopresis. During the appointment, the clinician will review strategies to increase continence by providing parent education on the following topics: how to collect and evaluate data on their child's bowel movements, how to establish and use a sit schedule, identifying behaviors that are precursors to bowel movements and how to use them to increase the probability of a bowel movement being continent, consequences for incontinence, and reinforcement for continence.
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study is comparing a multidisciplinary intervention for encopresis (MIE), consisting of both medical and behavioral components to treatment as usual control (TAU). Participants are first screened by a pediatric gastroenterologist and assessed and treated for any constipation or other potential medical complications. Following this, caregivers collect data on bowel movements and continence during a home baseline lasting no less than 14 days and no more than 21 days. Participants randomly assigned to treatment as usual or the treatment group, and begin attending daily appointments in clinic for 2 weeks. At appointments, the behavior team implements structured sits on the toilet to promote independent bowel movements (BMs). If an independent BM does not occur, the study team will administer a suppository to promote rapid release of the bowels and prompt the child to remain on the toilet following administration. In doing so, continent bowel movements are predictably evoked while the child is on the toilet, allowing for reinforcement with praise and preferred toys/activities. Eventually, suppositories are gradually decreased until the child is having BMs independently. Caregivers are trained to continue implementing the intervention following the clinic-based portion.

The purpose of the current study is to evaluate MIE using a large randomized clinical trial (RCT), addressing the Department of Defense Autism Research Program, Area of Interest of Therapies to Alleviate Conditions Co-Occurring with autism spectrum disorder (ASD). The researchers will recruit 112 children diagnosed with ASD, randomizing them to two weeks of MIE, or treatment as usual (TAU) consisting of behavioral consultation and medical intervention. This study will evaluate MIE compared to TAU and determine the optimal treatment length.

DETAILED DESCRIPTION:
Toilet training one's child is a nearly universal challenge for parents, but is a particularly distressing ordeal for parents of individuals with autism spectrum disorder (ASD). Whereas typically developing children generally stop having daytime toileting accidents (i.e., they achieve continence) by 2-4 years of age, most individuals with ASD are either delayed in their acquisition of toileting skills, or never achieve continence. Furthermore, toileting concerns are a significant contributor to the increased stress experienced by caregivers of those with ASD. Besides dramatically increasing their burden of care, not being fully toilet trained negatively impacts the individual with ASD's hygiene, self-confidence, physical comfort, and independence while also causing social stigma. Incontinence can also have serious collateral consequences, such as limiting exposure to important life experiences. Furthermore, without effective treatment these problems generally persist into adulthood.

One reason why strictly behavioral treatments of encopresis have shown only limited success may be due to the fact that it often has a medical etiology. Encopresis is when underwear are soiled by stool in children over the age of toilet training and long-standing constipation is the cause of encopresis in the majority of children who exhibit it. Children with ASD are more likely to have constipation than typically developing children. Constipation causes encopresis by creating a cycle of withholding bowel movements (withholding is the voluntary contraction of the external sphincter to avoid a bowel movement): constipation causes painful bowel movements, which triggers further withholding behavior, exacerbating constipation. Over time the colon adapts by dilating, which leads to larger fecal masses in the rectum. Thus, the passage of larger and harder (i.e., painful) stools further increases an individual's withholding behavior. Over time, the rectum and colon become so dilated that the individual loses sensation. With no urge to defecate, an individual is even more likely to have stool accumulate in the rectum and is also unable to control bowel movements. Looser stool may leak around hard stool leading to an unintended leakage and sometimes large evacuation of stool occurs without the individual realizing it.

Although purely medical approaches can successfully treat constipation in individuals with ASD, they have not shown long term success with encopresis. That is, medical approaches can treat a single episode of constipation, but without acquiring toileting skills, the individual is likely to become constipated again, repeating the cycle. Conversely, purely behavioral strategies have not been shown to be effective at treating encopresis in individuals with ASD, even when they are not experiencing constipation. One reason for this lack of success may have to do with the fact that it is often difficult to predict the timing of a bowel movement so that caregivers can ensure the individual is sitting on the toilet when one takes place and then reinforce continence. Thus, a multidisciplinary approach incorporating both medical and behavioral approaches is necessary in the treatment of encopresis in individuals with ASD.

This is an 8-week, randomized clinical trial of 112 children, ages 5 to 12 years, 11 months with ASD and encopresis. Participants will be randomized to receive either two weeks of MIE or one week of TAU. The study initially had a third study arm of one week of MIE treatment, which was discontinued in October of 2019.

ELIGIBILITY:
Inclusion Criteria:

* Males and females from 5 years of age to 12 years 11 months of age.
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of Autism Spectrum Disorder as established by clinical assessment, corroborated by the Autism Diagnostic Observational Schedule, Autism Diagnostic Interview-Revised and/or Childhood Autism Rating Scale-Second Edition.
* Fewer than 60% of days are continent days or more than 1 day out of 7 is an incontinent day over the previous 7 days (a continent day is defined as a day with at least one continent bowel movement. An incontinent day is a day with an incontinent bowel movement regardless of whether a continent bowel movement also occurs).
* Medication free or on stable medication (no changes in past 6 weeks and no planned changes for the next 6 months).
* Urine continent - Over half of the voids are continent when the child is with the parent and when the child is on a typical toileting routine.

Exclusion Criteria:

* Presence of a known medical condition in the child (based on medical history or physical examination) that would interfere with child's ability to control his/her anus. These include: history of any anal surgery, spinal dysraphism (e.g., spina bifida), other neurologic disorder affecting anal function, and prolonged/recurrent gastrointestinal infectious disease (e.g. Clostridium difficile colitis). In addition, the following may constitute exclusions following evaluation by a physician: inflammatory bowel disease, short gut syndrome, chronic diarrhea, or history of intestinal/abdominal surgery.
* Presence of a current serious behavioral problem or psychiatric condition that would require another treatment (e.g., psychotic disorder, major depression, moderate or greater aggression, severe disruptive behavior), based on information collected at screening and the Behavior Problems Inventory-01 (BPI-01).
* Currently receiving and caregiver refusal to discontinue ongoing behavioral or alternative medical intervention for encopresis.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Call, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Marcus Autism Center in Atlanta Georgia. Participant enrollment began October 25, 2017 and all study follow-up was complete by November 17, 2022.
Groups:
- Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week: Participants in this arm received the Multidisciplinary Intervention for Encopresis (MIE) for one week. MIE consists of daily clinic appointments, each of which lasts until a continent bowel movement occurs or 3 hours elapse. These participants discontinue the use of medication previously prescribed for the treatment of constipation, other than the suppositories used in the MIE treatment. During MIE, medical professionals resolve any constipation and oversee a regimen of over the counter medications that increase the predictability of a bowel movement. This study arm was discontinued in October 2019.
- Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks: Participants in this arm received the Multidisciplinary Intervention for Encopresis (MIE) for two weeks. MIE consists of daily clinic appointments, each of which lasts until a continent bowel movement occurs or 3 hours elapse. These participants discontinue the use of medication previously prescribed for the treatment of constipation, other than the suppositories used in the MIE treatment. During MIE, medical professionals resolve any constipation and oversee a regimen of over the counter medications that increase the predictability of a bowel movement.
- Treatment as Usual (TAU): Participants randomized to the Treatment as Usual (TAU) group continued to receive outpatient medical treatment of encopresis according to best practice guidelines by the pediatric gastroenterologist. In addition, participants in the TAU group received a 2-hour individual appointment in clinic with a doctoral level clinician with extensive experience in behavioral treatments for encopresis. During the appointment, the clinician reviewed strategies to increase continence by providing parent education on the following topics: how to collect and evaluate data on their child's bowel movements, how to establish and use a sit schedule, identifying behaviors that are precursors to bowel movements and how to use them to increase the probability of a bowel movement being continent, consequences for incontinence, and reinforcement for continence.
Period: Overall Study
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Started | 26 | 47 | 44
Completed | 18 | 32 | 40
Not Completed | 8 | 15 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 26 | 47 | 44 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.87 (1.61) | 7.38 (1.94) | 7.26 (1.69) | 7.12 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 8 | 26
  Male | 19 | 36 | 36 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 7 | 4 | 11
  Not Hispanic or Latino | 26 | 36 | 37 | 99
  Unknown or Not Reported | 0 | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 10 | 22 | 43
  Black or African American | 13 | 27 | 18 | 58
  Asian | 1 | 2 | 1 | 4
  More than one race or other race | 1 | 8 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 47 | 44 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Continent Bowel Movements
Description: The percentage to continent bowel movements, based on parent report during the prior 7 day period, are reported for Baseline and the end of treatment at Week 8.
Time Frame: Baseline, Week 8
Population: This analysis includes participants with complete data from parent reports of bowel movements during the prior week.
Measure: Mean (Standard Deviation); unit: percentage of bowel movements
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 37 | 40
percentage of bowel movements
  Baseline | 27.33 (29.72) | 16.99 (28.48) | 20.70 (25.80)
  Week 8: number analyzed (Participants) | 16 | 27 | 34
  Week 8 | 55.50 (33.18) | 79.69 (29.51) | 37.74 (35.92)

2. Secondary Outcome: Number of Children Responding to Treatment as Rated by the Clinical Global Impression Scale - Improvement (CGI-I) Score
Description: The Clinical Global Impression Scale - Improvement (CGI-I) is a single item asking clinicians to indicate the degree of improvement following treatment on a 7-point scale. Responses are 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. This study is interested in the proportion of children who are rated by the Independent Evaluator as "Much Improved" or "Very Much Improved" on the CGI-I at Week 8. Responding to treatment is defined as a score of 1 or 2, while scores of 3 to 7 are considered as not responding to treatment. Response to treatment is analyzed through imputation, consistent with an intent to treat approach, where participants who withdrew from the study or were lost to follow-up prior to the Week 8 assessment are considered to be non-responders.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 47 | 44
Participants
  No response (CGI-I score of 3 to 7) | 16 | 26 | 37
  Response (CGI-I score of 1 or 2) | 10 | 21 | 7

3. Secondary Outcome: Parenting Stress Index Short Form Total Score
Description: The Parenting Stress Index Short Form (PSI-SF) is a 36-item questionnaire assessing parental stress. It has three subscales of Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Each subscale has 12 items where responses are given on a 5-point scale where 1 = strongly disagree and 5 = strongly agree. Scores for subscales range from 12 to 60 and the total score ranges from 36 to 180. Higher scores indicate greater parental stress.
Time Frame: Baseline, Week 8
Population: This analysis includes parents of children who were participating in the study at the indicated study visit. Twenty-seven participants withdrew or were lost to follow-up prior to the Week 8 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 47 | 44
score on a scale
  Baseline | 82.38 (23.25) | 81.72 (24.79) | 91.22 (20.94)
  Week 8: number analyzed (Participants) | 18 | 32 | 40
  Week 8 | 80.88 (23.95) | 82.76 (29.68) | 89.19 (24.45)

4. Secondary Outcome: Caregiver Strain Questionnaire - Short Form 7 (CGSQ-SF7) Objective Strain Subscale Score
Description: The Caregiver Strain Questionnaire - Short Form (CGSQ-SF7) assesses parental stress and strain in the prior month in caregivers who are caring for a child with behavioral disorders. The CGSQ-SF includes 7 items where responses are given on a 5-point scale where "not at all" is scored as 0 and "very much" is scored as 4. The CGSQ-SF7 has two subscales: Objective Strain with four items, and Subjective Internalized Strain with three items. The total score for the Objective Strain subscale ranges from 0 to 16 and higher scores indicate greater parental strain.
Time Frame: Baseline, Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 47 | 44
score on a scale
  Baseline Objective Strain Subscale Score | 9.68 (4.35) | 9.86 (4.51) | 9.40 (3.91)
  Week 8 Objective Strain Subscale Score: number analyzed (Participants) | 18 | 32 | 40
  Week 8 Objective Strain Subscale Score | 9.53 (3.41) | 8.21 (4.20) | 9.29 (4.04)

5. Secondary Outcome: Caregiver Strain Questionnaire - Short Form 7 (CGSQ-SF7) Subjective Internalized Strain Subscale Score
Description: The Caregiver Strain Questionnaire - Short Form (CGSQ-SF7) assesses parental stress and strain in the prior month in caregivers who are caring for a child with behavioral disorders. The CGSQ-SF includes 7 items where responses are given on a 5-point scale where "not at all" is scored as 0 and "very much" is scored as 4. The CGSQ-SF7 has two subscales: Objective Strain with four items, and Subjective Internalized Strain with three items. The total score for the Subjective Internalized Strain subscale ranges from 0 to 12 and higher scores indicate greater parental strain.
Time Frame: Baseline, Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 47 | 44
score on a scale
  Baseline Subjective Internalized Strain Subscale Score | 8.88 (3.26) | 10.16 (3.89) | 9.29 (3.06)
  Week 8 Subjective Internalized Strain Subscale Score: number analyzed (Participants) | 18 | 32 | 40
  Week 8 Subjective Internalized Strain Subscale Score | 9.06 (3.13) | 7.24 (3.51) | 9.58 (3.58)

6. Secondary Outcome: Caregiver Strain Questionnaire - Short Form (CGSQ-SF7) Total Score
Description: The Caregiver Strain Questionnaire - Short Form (CGSQ-SF7) assesses parental stress and strain in the prior month in caregivers who are caring for a child with behavioral disorders. The CGSQ-SF includes 7 items where responses are given on a 5-point scale where "not at all" is scored as 0 and "very much" is scored as 4. The CGSQ-SF7 has two subscales: Objective Strain with four items, and Subjective Internalized Strain with three items. A total score is obtained by adding the scores for each subscale. Total scores range from 0 to 28 where higher scores indicate greater caregiver strain.
Time Frame: Baseline, Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
Number analyzed (Participants) | 26 | 47 | 44
score on a scale
  Baseline | 18.56 (7.12) | 20.03 (7.58) | 18.69 (6.46)
  Week 8: number analyzed (Participants) | 18 | 32 | 40
  Week 8 | 18.59 (6.15) | 15.45 (7.30) | 18.87 (7.05)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of the baseline visit through the follow-up assessment at Week 8.
Arm/Group | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/47 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/47 | 0/44
Other Adverse Events (participants affected / at risk) | 24/26 | 35/47 | 41/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multidisciplinary Intervention for Encopresis (MIE) Treatment for One Week (N=26) | Multidisciplinary Intervention for Encopresis (MIE) Treatment for Two Weeks (N=47) | Treatment as Usual (TAU) (N=44)
Seizures (Nervous system disorders) | 0 | 1 | 0
Ear infection (Ear and labyrinth disorders) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 5 | 4 | 4
Sore throat (General disorders) | 1 | 0 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 3
Constipation (Gastrointestinal disorders) | 3 | 14 | 8
Excessive appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 0 | 1 | 0
Tired during the day (General disorders) | 0 | 1 | 0
Difficulty falling asleep (General disorders) | 3 | 1 | 5
Early morning waking (General disorders) | 3 | 0 | 0
Interrupted sleep (General disorders) | 0 | 0 | 1
Fever (Infections and infestations) | 1 | 0 | 2
Allergies (Immune system disorders) | 1 | 2 | 0
Swollen tonsils (Infections and infestations) | 1 | 0 | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Difficulty staying asleep (General disorders) | 1 | 1 | 2
Red itchy rash on leg (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ear bleed (Ear and labyrinth disorders) | 0 | 1 | 0
Abrasion on chin (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bump on back of head (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cavity (General disorders) | 0 | 0 | 1
Cut on ear from haircut (Injury, poisoning and procedural complications) | 0 | 0 | 1
Problem behavior (General disorders) | 0 | 1 | 0
Mid-sleep awakening (General disorders) | 0 | 2 | 2
Inappropriate language (General disorders) | 0 | 1 | 0
Difficulty waking up (General disorders) | 0 | 0 | 2
Strep throat (Infections and infestations) | 0 | 0 | 1
Infected toe nail (Infections and infestations) | 0 | 0 | 1
Naps during the day (General disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03197922/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03197922/ICF_000.pdf